CLINICAL TRIAL: NCT03810586
Title: Comparison of Continuous Blood Pressure Measurement Using a Non-invasive Photo Plethysmography-based Monitor With the Gold Standard Sphygmomanometer-based Holter Monitor
Brief Title: Comparing PPG-based Blood Pressure Measurement to the Gold Standard Manometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biobeat Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biobeat002
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hypertension; Blood Pressure Disorders
Keywords: Hypertension; Continuous Monitoring; Non-invasive Blood Pressure; Non-invasive Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Recruitment will be via printed advertisements distributed throughout the medical center. Volunteers will arrive on the morning of the test and fill a questionnaire about their demographics and every day activities. After completing the questionnaire, the participants will be connected to both devices, one on each arm and undergo a briefing about both devices. A first calibration measurement will take place followed by BP measurement every 20 minutes, and up to a 24 hour period. After 24 hours of measurements, the participants will return to Hadassah Medical Center and fill in another questionnaire, which will include feedback on the use of both devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparing blood pressure measurement (Experimental): In each volunteer, non-invasive measurements of blood pressure will be taken at the same time using a holter manometry device (HUGECARE NIBP Monitor) and the Biobeat BB-613 device, and compared, to show the accuracy and the comparability of the BB-613. As mentioned in the protocol, there would be no medical interventions within the scope of this study. In case hypertension will be observed in a volunteer, the volunteer will be advised by the investigators to see his physician for further evaluation.
  Interventions: Device: Non-invasive measurement of blood pressure

INTERVENTIONS:
Device: Non-invasive measurement of blood pressure — Comparing non-invasive measurement of blood pressure using the PPG-based BB-613 device to a blood pressure manomtry holter device (HUGECARE NIBP Monitor)

SUMMARY:
Continuous blood pressure (BP) measurement is in use today with an ambulatory, sphygmomanometer-based, device. This device, also called BP Holter, gives essential data for the clinician, allowing better hypertension (HTN) diagnosis and treatment. Alongside, the device has some substantial limitations preventing its use as a longer term BP monitoring allowing better HTN control. A new method of continuous BP monitoring, based on photo plethysmography (PPG), has been invented to ease patients' use and increase their responsiveness. This study aims to check whether the new, PPG-based method, of BP measurement can be as good as the current, gold standard, sphygmomanometer-based device.

DETAILED DESCRIPTION:
HTN is a major risk factor for cerebrovascular morbidity and mortality, yet its identification can be delayed due to lack of overt symptoms, relying on BP measurements for diagnosis. Several BP monitoring techniques are used in clinics and hospitals, and there is also an outpatient method that is used for 24-hour BP monitoring, based on a sphygmomanometer. The general notion is that by using tight BP monitoring in the clinic and during the day, the health system will be able to diagnose hypertension among individuals at an early stage, including high risk patients in the community.

Ambulatory BP monitoring for a period of 24 hours is considered to be better than measurements taken in a clinic setting. First, 24 hours monitoring performed at home can help confirm that hypertension actually does exist, thus ruling out the potential of "white coat syndrome". Second, measurements of BP during sleep also have a predictive value for hypertension in high risk patients. Furthermore, ambulatory BP measurements are a stronger predictor of all-cause and cardiovascular mortality than BP measurements in the clinic. Finally, continuous BP monitoring is beneficial for controlling hypertension in diagnosed and treated patients.

The gold standard ambulatory non-invasive BP monitor that is in broad use today is a sphygmomanometer-based device that includes a cuff, which contracts around the patient's arm and measures BP every 15 to 20 minutes. The cuff is usually uncomfortable for the patients and could prevent them from doing their everyday activities. It can also disrupt the quality of their sleep at night. For these reasons patients are sometimes reluctant to use it. A more comfortable, user- friendly device, which allows a non-invasive, continuous BP measurement will provide a simple, more efficient way for BP monitoring, and will potentially enable to improve the outcome of medical treatment.

A new way for continuous non-invasive BP monitoring is based on the reflective photo plethysmography (PPG) method. A company called "Biobeat" invented a device that measures PPG wave in high temporal resolution that maintains more properties and markings of the original pulse wave than usual PPG-based devices, thereby enabling to provide data on several physiological parameters other than Heart Rate (HR) and blood oxygen saturation, such as: Systolic Blood Pressure (SBP) and its variation, Diastolic Blood Pressure (DBP) and its variation, Pulse Pressure and more. This device can also send and surveillance. The Biobeat device (BB-613) includes either a wearable watch or a patch with a sticker that the patient puts on his/her body. This device may increase the patient's willingness to use it and can also make the measurement more reliable (explanation on the PPG-based sensor and the device itself are provided in the appendixes).

The measurements are transferred via Wi-Fi to the patient's doctor and allows close monitoring.

The purpose of the study The study's main purpose is to compare continuous 24-hour BP measurement using the non-invasive PPG-based BB-613 device with one of the gold standard sphygmomanometer-based devices that is currently-used throughout the Israeli health system (HUGECARE NIBP Monitor). As accepted according to the AAMI (Association for the Advancement of Medical Instrumentation) and the European Hypertension Society, the parameters that are investigated in this study will be systolic BP, diastolic BP and the average between them (MAP).

The use of the PPG sensor for BP measurement will be considered as successful if there will be correlation of at least 5/10/15 mmHg between the measurements of both the PPG sensor and the sphygmomanometer-based Holter. The difference between measurements of the PPG and manometer devices will be less than 5 mmHg in at least 75% of the measurements, less than 10 mmHg in at least 90% of the measurements and less than 15 mmHg in at least 96% of the measurements. The results will fulfil at least two of these criteria.

In addition to the BP measurement comparison, in this study the investigators will also compare the degree of comfort and accessibility for participants between the Bio Beat device and the gold standard Holter device that is currently in use.

Study hypothesis The study's hypothesis is that the PPG-based sensor will give reliable results of continuous BP monitoring in a comfortable and user-friendly way. In addition, the accuracy of the sensor will not be inferior to the Holter that is now in use.

ELIGIBILITY:
Inclusion Criteria:

* Either healthy or chronically ill who are treated accordingly and with no need of any medical intervention during the study.

Exclusion Criteria:

* A volunteer's refusal to enter the study.
* Patients who are currently in hospitalization or in medical assessment.
* Pregnant women and children under 18.
* Volunteers with powerless jurisdiction.
* Workers of the Hadassah Medical Center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Accurate and comparable blood pressure measurement by BB-613 | 24 hours per participant
  Blood pressure measurements using the PPG-based BB-613 device will be taken and compared to blood pressure measurements taken at the same time using the holter device HUGECARE NIBP Monitor, with the aim of showing they are comparable

CONTACTS AND LOCATIONS:
Overall Officials: Dean Nachman, MD, Principal Investigator — The Hadassah Ein Kerem Medical Center, Jerusalem
Locations (1):
- The Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nachman D, Gilan A, Goldstein N, Constantini K, Littman R, Eisenkraft A, Grossman E, Gepner Y. Twenty-Four-Hour Ambulatory Blood Pressure Measurement Using a Novel Noninvasive, Cuffless, Wireless Device. Am J Hypertens. 2021 Nov 20;34(11):1171-1180. doi: 10.1093/ajh/hpab095. PMID 34143867